CLINICAL TRIAL: NCT04960228
Title: Enhancing COVID-19 Vaccination Intentions by Eliciting Prosocial Altruistic Motives: Evaluating the Efficacy of a Brief Video-Based Intervention
Brief Title: Exploring Changes in COVID-19 Vaccination Intentions by Prompting Altruistic Motives Using a Video Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeev Rosberger (Other)
Responsible Party: Sponsor-Investigator, Zeev Rosberger, Senior Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-2877
Record Dates: First submitted 2021-06-30; First posted 2021-07-13 (Actual); Results first posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Vaccine Refusal
Keywords: Vaccine Hesitancy; Vaccine Decision Making; COVID-19
MeSH Terms: conditions — Vaccination Refusal; Vaccination Hesitancy; COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either the video intervention or informational text control condition using a 1:1 randomization ratio.
Who Masked: Investigator
Masking Description: All data collection and group assignment will be conducted by the survey company, Dynata. Participants' intervention group assignments will be unavailable to the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Altruism Video Intervention (Experimental): Participants will watch a 3-minute video about COVID-19 vaccination that elicits altruistic motives. The role of this arm is to test whether altruistic themes are an effective way to promote COVID-19 vaccination amongst young people and whether a video format is preferable for this group.
  Interventions: Behavioral: Altruism Video
- Informational Text Intervention (Active Comparator): Participants will read a brief informational text including information drawn from the Public Health Agency of Canada website (https://www.canada.ca/en/public-health/services/diseases/2019-novel-coronavirus-infection/prevention-risks.html#self). The purpose of this arm is to provide an active comparator with information about COVID-19 preventative health behaviors that has been strongly recommended to the public since the beginning of the pandemic. By doing this, we will assess if the video intervention changes vaccination intentions more than a presentation of general, well-known COVID-19 related information.
  Interventions: Behavioral: COVID-19 Informational Text

INTERVENTIONS:
Behavioral: Altruism Video — The video provides three vignettes about a diverse set of people who may be more vulnerable to serious health consequences from COVID-19. In each of the stories, high vaccine uptake of those around these vulnerable individuals serves to protect them. This communicates that getting the COVID-19 vaccine can be done for prosocial reasons and to foster a sense of community, as it provides protection not only to oneself, but also to others.
  Arms: Altruism Video Intervention
Behavioral: COVID-19 Informational Text — The topics included in the text are how COVID-19 spreads, hygiene, physical distancing, and travel restrictions. Participants will complete three comprehension questions, one after each of the following sections: hygiene, physical distancing, and travel restrictions.
  Arms: Informational Text Intervention

SUMMARY:
As Canada records over 1,400,000 COVID-19 infections and 26,000 deaths, the need to stop the spread of the virus has become increasingly critical. Although younger individuals (aged 20-39) have lower hospitalisation and death rates than older adults, they have high rates of infection and may be less willing to accept a vaccine because they consider the disease to be less dangerous for themselves. It is of concern that around 30% of Canadians, especially younger adults, will not be willing to accept a COVID-19 vaccine. Vaccination will be the best method to control the pandemic in the future and protect those at higher risk of hospitalisation and death (e.g., elderly, those with chronic diseases). Therefore, achieving high rates of vaccination coverage among younger adults is very important in the long run to protect not only themselves but also others. For the experimental condition, the investigators will develop a brief video that will promote the vaccine's protection of others (altruism). For the control condition, the investigators will create an informational text on COVID-19 preventative health measures based on recommendations from the Public Health Agency of Canada. 2630 younger adults (aged 20 to 39) who have not yet received a dose of a COVID-19 vaccine will be recruited. To match Canadian demographics, participants will be recruited using the following quotas to reflect census data from Statistics Canada: 50% male and 50% female; 80% Anglophone and 20% Francophone; 80% urban and 20% rural; and 50% household income level less than $75,000 and 50% household income greater than $75,000. Half of the participants will be randomly assigned to watch the video, with the other half reading the text. In both groups, participants will complete a short online survey before and after viewing the video or reading the text. The goal is to assess the efficacy of the video on increasing younger adults' willingness to get a COVID-19 vaccine. The research team is partnering in this study with key agencies, e.g., Public Health Agency of Canada (PHAC), National Advisory Committee on Immunization (NACI), and the Institut National de Santé Publique du Québec (INSPQ) to help communicate the research findings to the general population.

DETAILED DESCRIPTION:
The COVID-19 vaccine is the most effective way to arrest the pandemic. A high vaccine acceptance rate is needed to achieve community immunity; however, current COVID-19 vaccine acceptance rate remains low, particularly among younger Canadians. There have been no studies that have examined the impact of altruism on COVID-19 vaccine intentions using a video-based intervention. The investigators will examine the efficacy of a video intervention eliciting altruism on increasing younger Canadians' (ages 20-39) intentions to receive the COVID-19 vaccine using a randomized control trial. The results of this study will be used by public health authorities to increase COVID-19 vaccine uptake. There are two objectives of the study: 1) to assess the within-participant efficacy of the video intervention in increasing vaccine intentions; 2) to assess the between-participant efficacy of the video intervention in increasing vaccine intentions.

A 10-minute survey will be administered online to a sample of 2630 Canadian residents aged 20-39 years old and is available in both English and French. To calculate the required sample size for the within-participant change in vaccine hesitancy (i.e., pre-post video intervention) the investigators used survey data showing that approximately 40% of Canadians in this age group are COVID-19 vaccine hesitant i.e., don't know yet or would refuse vaccination. Estimating a 5% decrease of hesitancy in the video intervention group and a correlation of about 0.45 between paired observations, this group requires a sample size of 1315 pairs for detecting a 5% change of marginal proportions at a power of 80% and two-sided significance of 5%.

Participants will be randomized using a one-to-one ratio. Thus, 50% will be allocated to the video intervention and 50% to the text intervention. Using equal size groups will allow for the detection of a between group difference in vaccine intentions of 5-6% with a power of 0.8 and a two-sided significance of 5%. The total sample required for this study is 2630 participants i.e., 1315 in the video intervention group and 1315 in the text intervention group.

The investigators have contracted Dynata, the world's largest first-party data and insight platform, to conduct recruitment and host the survey. Dynata will send invitations in various forms (e.g., e-mail invitations, text messages and in-app alerts) to recruit eligible participants from their existing panel (individuals who have signed with Dynata and have expressed willingness to receive invitations to various appropriate surveys) until recruitment goals and quotas are met.

Stratified randomization will be used to allocate participants to either: 1) video intervention: viewing a 2-minute altruism-eliciting video, or 2) text intervention: reading a text containing information from the Public Health Agency of Canada about general health behaviours and public health recommendations concerning COVID-19, e.g., hand hygiene and respiratory etiquette, wearing non-medical masks, physical distancing, etc. Within each stratum (first language, sex, population density and household income), participants will be allocated randomly using a one-to-one ratio (one to the video intervention and one to the text intervention).

Participants will first be asked to answer several socio-demographic questions and will be asked to choose one of the following categories which describe their COVID-19 vaccine decision-making stage according to the Precaution Adoption Process Model (PAPM): unengaged, undecided, decided not to receive the vaccine, or decided to receive the vaccine. Subsequently, depending on their randomly assigned condition, participants will either be shown a 2-minute altruism-eliciting video, or a brief informational text. After viewing this content, to ensure that participants paid attention, participants will answer questions about the contents to check their understanding. Finally, participants will: 1) once again be asked to choose their COVID-19 vaccine decision-making stage; 2) be asked questions regarding previous vaccination history (e.g., seasonal influenza), lifestyle factors, self-perceived health status, personal history of SARS-CoV-2 infection, and preferred health-information channels; and 3) complete validated scales regarding altruism, empathy, personal distress, and vaccine hesitancy.

To test the outcome for objective 1, the McNemar's test will be used to compare paired (pre-post video intervention) proportions. To control for the potential effect of other factors (e.g., sociodemographics, previous influenza vaccination, lifestyle factors), the investigators will conduct multivariate analyses (General Estimating Equations) and estimate the associations between these factors and changes in COVID-19 vaccine intentions. For objective 2, the difference in proportions between the video intervention and text intervention will be analyzed using the Chi-square test. The investigators will test for significant differences in predictor variables between the two groups and use logistic regression analyses to estimate the associations between these variables and the outcome (vaccine acceptability). The significance level will be set at α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Residing within Canada and aged between 20 and 39 years.

Exclusion Criteria:

* Having received at least one dose of a COVID-19 vaccine

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2097 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Rosberger, PhD, Principal Investigator — Lady Davis Institute for Medical Research of the Jewish General Hospital
Locations (1):
- Lady Davis Insitutute for Medical Research, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Consent form, data collection method, and organizational policy means only aggregated data will be shared with other researchers.

REFERENCES:
- [Background] Li M, Taylor EG, Atkins KE, Chapman GB, Galvani AP. Stimulating Influenza Vaccination via Prosocial Motives. PLoS One. 2016 Jul 26;11(7):e0159780. doi: 10.1371/journal.pone.0159780. eCollection 2016. PMID 27459237
- [Background] Brewer NT, Chapman GB, Rothman AJ, Leask J, Kempe A. Increasing Vaccination: Putting Psychological Science Into Action. Psychol Sci Public Interest. 2017 Dec;18(3):149-207. doi: 10.1177/1529100618760521. PMID 29611455
- [Background] Rieger M. Triggering altruism increases the willingness to get vaccinated against COVID- 19. Social Health and Behavior. 2020; 3(3): 78.
- [Derived] Zhu P, Tatar O, Griffin-Mathieu G, Perez S, Haward B, Zimet G, Tunis M, Dube E, Rosberger Z. The Efficacy of a Brief, Altruism-Eliciting Video Intervention in Enhancing COVID-19 Vaccination Intentions Among a Population-Based Sample of Younger Adults: Randomized Controlled Trial. JMIR Public Health Surveill. 2022 May 30;8(5):e37328. doi: 10.2196/37328. PMID 35544437
- See also: Recent poll detailing levels of vaccine hesitancy among Canadians, including young Canadians. — http://www.ipsos.com/en-ca/news-polls/Eight-in-Ten-Canadians-Vaccinated-Remaining-Need-Convinced
- See also: Summary of COVID-19 statistics in Canada — https://health-infobase.canada.ca/covid-19/epidemiological-summary-covid-19-cases.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from July 30th to September 13th, 2021. All recruitment took place online through the survey company Dynata.
Pre-assignment Details: 14,298 participants began the survey. Exclusion occurred during a screening item to ensure participants audio/video (1396 excluded) was working for the study, and by assessing inclusion/exclusion criteria (9752 excluded). Additionally, 238 participants did not consent to participate, and 815 dropped out before randomization.
Period: Overall Study
Arm/Group | Altruism Video Intervention | Informational Text Intervention
Started (Randomized to intervention) | 1098 | 999
Completed (Completed full survey including post-intervention outcome measure) | 810 | 813
Not Completed | 288 | 186
Not completed — Withdrawal by Subject | 216 | 35
Not completed — Failed attention check | 69 | 148
Not completed — Flagged for response quality by Dynata | 3 | 3

BASELINE CHARACTERISTICS:
Population: The number analyzed were those who completed the full survey, passed the in-survey attention checks, and were retained during post-hoc data cleaning methods (outlying survey response times, straight-lined responses).
Groups:
- Total: Total of all reporting groups
Arm/Group | Altruism Video Intervention | Informational Text Intervention | Total
Number analyzed (Participants) | 686 | 687 | 1373
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed were those who completed the full survey, passed the in-survey attention checks, and were retained during post-hoc data cleaning methods (outlying survey response times, straight-lined responses).
  years | 30.7 (5.4) | 30.7 (5.3) | 30.7 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Male/Female biological sex. Population: The number analyzed were those who completed the full survey, passed the in-survey attention checks, and were retained during post-hoc data cleaning methods (outlying survey response times, straight-lined responses).
  Participants
    Female | 370 | 370 | 740
    Male | 316 | 317 | 633
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Categories for ethnicity recommended by Statistics Canada. These categories were chosen to facilitate interpretation by public health agencies in Canada. Population: The number analyzed were those who completed the full survey, passed the in-survey attention checks, and were retained during post-hoc data cleaning methods (outlying survey response times, straight-lined responses).
  Participants
    Ethnicity (Statistics Canada): North American Aboriginal (e.g., First Nations, Inuit, Metis) | 62 | 45 | 107
    Ethnicity (Statistics Canada): Other North American (e.g., Canadian, American, Ontarian, Quebecois, Acadian) | 301 | 331 | 632
    Ethnicity (Statistics Canada): European (e.g., British, French, Western European, Eastern European) | 158 | 156 | 314
    Ethnicity (Statistics Canada): Caribbean (e.g., Cuban, Haitian, Jamaican) | 33 | 23 | 56
    Ethnicity (Statistics Canada): Latin, Central and South American (e.g., Mexican, Argentinian, Brazilian, Chilean) | 16 | 14 | 30
    Ethnicity (Statistics Canada): African (e.g., Central and West African, North African, Southern Africa) | 30 | 30 | 60
    Ethnicity (Statistics Canada): Asian (e.g., West Central Asian, South Asian, East and Southeast Asian) | 42 | 42 | 84
    Ethnicity (Statistics Canada): Oceania (e.g., Australian, New Zealander, Pacific Islander) | 0 | 2 | 2
    Ethnicity (Statistics Canada): Other (free response) | 44 | 44 | 88
Region of Enrollment [Count of Participants; unit: Participants] — Province or Territory of residence Population: The number analyzed were those who completed the full survey, passed the in-survey attention checks, and were retained during post-hoc data cleaning methods (outlying survey response times, straight-lined responses).
  Participants
    Canada: Alberta | 106 | 105 | 211
    Canada: British Columbia | 67 | 70 | 137
    Canada: Manitoba | 33 | 27 | 60
    Canada: New Brunswick | 10 | 22 | 32
    Canada: Newfoundland and Labrador | 14 | 17 | 31
    Canada: Nova Scotia | 14 | 22 | 36
    Canada: Nunavet | 1 | 2 | 3
    Canada: Ontario | 376 | 345 | 721
    Canada: Prince Edward Island | 2 | 4 | 6
    Canada: Quebec | 43 | 49 | 92
    Canada: Saskatchewan | 19 | 24 | 43
    Canada: Yukon | 1 | 0 | 1
COVID-19 Vaccine Intentions Pre-Intervention [Count of Participants; unit: Participants] — Vaccine intentions are measured using one item: "Which of the following best describes your thoughts about a COVID-19 vaccine?". Participants will then indicate their vaccine intention stage, adapted from the Precaution Adoption Process Model (PAPM): I have not thought about receiving the COVID-19 vaccine, I am undecided about receiving the COVID-19 vaccine, I do not want to receive the COVID-19 vaccine, and I do want to receive the COVID-19 vaccine. Participants will answer this item before (pre) and after (post) the intervention has been administered, all within the same survey.
  Participants
    Unengaged | 74 | 73 | 147
    Undecided | 234 | 255 | 489
    Decided Not | 292 | 272 | 564
    Decided To | 86 | 87 | 173

OUTCOME MEASURES:

1. Primary Outcome: Post Intervention Vaccine Intentions
Description: Vaccine intentions are measured using one item: "Which of the following best describes your thoughts about a COVID-19 vaccine?". Participants will then indicate their vaccine intention stage, adapted from the Precaution Adoption Process Model (PAPM): I have not thought about receiving the COVID-19 vaccine, I am undecided about receiving the COVID-19 vaccine, I do not want to receive the COVID-19 vaccine, and I do want to receive the COVID-19 vaccine. Participants will answer this item before (pre) and after (post) the intervention has been administered, all within the same survey.
Time Frame: Pre-post intervention, within the same survey. The length of the survey is projected to be about 10 minutes.
Population: Canadian residents aged 20-39 who had not received any dose of a COVID-19 vaccine at the time of recruitment.
Measure: Count of Participants; unit: Participants
Arm/Group | Altruism Video Intervention | Informational Text Intervention
Number analyzed (Participants) | 686 | 687
Participants
  Unengaged | 54 | 47
  Undecided | 236 | 249
  Decided Not | 277 | 285
  Decided To | 119 | 106

ADVERSE EVENTS:
Time Frame: Adverse data information was only collected during the administered survey (10-15 minutes length) within the recruitment period (July 30th, 2021 - September 13th, 2021).
Description: Adverse event collection was provided to us by the survey fielding company, Dynata.
Arm/Group | Altruism Video Intervention | Informational Text Intervention
All-Cause Mortality (participants affected / at risk) | 0/1098 | 0/999
Serious Adverse Events (participants affected / at risk) | 0/1098 | 0/999
Other Adverse Events (participants affected / at risk) | 0/1098 | 0/999

LIMITATIONS AND CAVEATS:
Several limitations presented themselves during study recruitment. COVID-19 vaccination rates amongst our target population (Canadian young adults) increased significantly, especially driven by vaccination mandates that were introduced in several provinces. This meant we were not able to reach our target sample size (2630 participants), preventing adequate power for calculations and the filling of our pre-specified sample quotas (limiting generalizability). Additional, we used self-reported data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT04960228/Prot_002.pdf
  • Statistical Analysis Plan (2022-02-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT04960228/SAP_003.pdf
  • Informed Consent Form: English Version (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT04960228/ICF_004.pdf